CLINICAL TRIAL: NCT02092272
Title: Does Providing Instructional Exercise Videos Increase Patient Adherence Compared to In-office Instruction by Physician When Using Eccentric Exercises to Treat Shoulder Pain in Adults?
Brief Title: Eccentric Exercises for Shoulder Pain
Acronym: Eccentric
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the PI left our facility and the new staff prefer alternate excersises
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FWH20140038H
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- instructional exercise video source (Experimental): instructional exercise video source
  Interventions: Behavioral: instructional exercise video source
- Standard Therapy (No Intervention): Standard Therapy

INTERVENTIONS:
Behavioral: instructional exercise video source — instructional exercise video source
  Arms: instructional exercise video source

SUMMARY:
Patients will be randomly assigned to one of two groups using a random number generator. Group 1 will be provided with in-office instruction of standard of care eccentric exercises for rotator cuff tendinopathy. Group 2 will be provided with in-office instruction as well as a instructional exercise video source (DVD) to take home as a reminder on how to perform two specific standard of care eccentric exercises for rotator cuff tendinopathy. Each group will be given a card to track adherence to the standard of care eccentric exercise routine as measured only by the days that they accomplish their exercises. Study exercise diary will be collected after 12 weeks of treatment. Eccentric exercises are taught as part of standard of care for rotator cuff tendinopathy.

DETAILED DESCRIPTION:
DoD beneficiaries age 18 or older will be recruited from the clinics at the Mike O'Callaghan Federal Medical Center (MOFMC). Subjects meeting the inclusion/exclusion criteria will be offered an opportunity to participate:

Screening Visit:

* Obtain signed Informed Consent Document and HIPAA Authorization.
* Verify inclusion/exclusion criteria

Visit 1 (may occur same day as Screening Visit):

* Subjects will be randomly assigned to one of two groups by the Research Coordinator using a random number generator, thus the Investigators will be blinded to the group assignments:

  * Group 1: in-office instruction of the standard of care eccentric exercise regimen for rotator cuff tendinopathy.
  * Group 2: in-office instruction of the standard of care eccentric exercise regimen for rotator cuff tendinopathy and an instructional exercise video source (DVD).
* Subjects will be given a study exercise diary to track adherence to the standard of care eccentric exercise routine.

Visit 2 (12 weeks post Visit 1):

• Study exercise diary will be collected to assess adherence. If the subject is unable to come in, they can return the study exercise diary via mail, or electronic mail.

ELIGIBILITY:
Inclusion:

* DoD beneficiary patient 18 years or older
* Diagnosis of chronic (>30 days) shoulder pain of any etiology (traumatic vs over-use injury)

Exclusion:

* Patients < 18 years of age
* Patients with acute injury (fracture or injury within 30 days)
* Patients unable to accomplish eccentric exercise regimen without assistance
* Patients unable to view DVD
* Pregnant women
* Patients unable to read and/or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
patient adherence to standard of care eccentric exercise regimens | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Connor McKeown, MD, Principal Investigator — Mike O'Callaghan Military Hospital
Locations (1):
- Mike O'Callaghan Federal Hospital, Nellis Air Force Base, Nevada, United States